CLINICAL TRIAL: NCT02332070
Title: Timing of Coronary Angiography and Multivariate Risk for Cardiac Surgery Associated Acute Kidney Injury and Major Adverse Renal and Cardiac Events (MARCE)
Brief Title: Timing of Coronary Angiography, Cardiac Surgery, and Adverse Renal and Cardiac Events (MARCE)
Acronym: MARCE
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 014-096
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Acute Kidney Injury; Renal Insufficiency
Keywords: acute kidney injury; coronary angiography; cardiac surgery; adverse events; iodinated contrast; Thoracic Surgery
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cardiac surgery — coronary artery bypass surgery and or cardiac valve surgery with cardiopulmonary bypass

SUMMARY:
1. To examine two main predictor variables independently and then jointly in stratified and multivariate analyses for the outcomes of CSA-AKI, MARCE, need for RRT, and inpatient mortality, and the composite, as well as the outcomes of 30 day rehospitalization or death, and finally for the days out of hospital and alive adjusted to person-year of time

   1. Days from coronary angiogram performed with IOCM to cardiac surgery (1, 2, 3, etc)
   2. Thakar Acute Renal Failure (ARF) score (1 to 17)
2. To examine the interrelationships between time in days between angiogram and surgery and the ARF Score with the Society of Thoracic Surgery (STS) Risk score for mortality

DETAILED DESCRIPTION:
Background: Despite advances in cardiac surgical techniques, modern anesthesia, and adjunctive medical therapies, cardiac-surgery associated acute kidney injury (CSA-AKI) remains a frequent and important complication. With advancing age and more severe comorbidities present in patients undergoing cardiac surgery, multivariate scores (e.g. Thakar Acute Renal Failure [ARF] score) would anticipate future higher rates of CSA-AKI that resolve, lead to progressive chronic kidney disease (CKD), require renal replacement therapy (RRT), and are associated major adverse cardiac events with early and later mortality. Mehta and colleagues in a study of 2441 cases suggested that CSA-AKI was associated with the time between the diagnostic coronary angiogram and the subsequent surgery. This suggested that superimposed risk of contrast-induced AKI (CI-AKI) followed by cardiac surgery was a serial insult to the kidneys producing the clinical syndrome of CSA-AKI. However, Andersen and coworkers, in a study of 285 consecutive patients concluded that cardiac surgery within 1-3 days of coronary angiography was safe and not associated with CSA-AKI. Attempts at evaluating CSA-AKI risk prediction models have been limited by small sample sizes. For example, Kiers et el attempted to evaluate 8 CSA-AKI risk models in 1388 patients and found several scores could not be computed due to lack of information and those that could have unstable point estimates for C-statistics and other measures. As a result, CSA-AKI risk scores and attempts to improve quality of care have not been applied in a widespread manner to cardiac surgical cases. Thus we propose to evaluate these key concepts in a large dataset which captures important clinical events such as CI-AKI and type of contrast used followed by CSA-AKI and associated major adverse renal and cardiac events (MARCE) including the need for RRT, myocardial infarction, stroke, heart failure, hospitalizations (cardiac or renal) and death. We aim to derive a practical approach in determining the optimal waiting period from the time of angiography to cardiac surgery according to risk for CSA-AKI in subjects who have received iso-osmolar contrast media (IOCM) with preoperative angiography, as that agent has been shown to have the lowest risk of CI-AKI.

Specific Aims:

1. To examine two main predictor variables independently and then jointly in stratified and multivariate analyses for the outcomes of CSA-AKI, MARCE, need for RRT, and inpatient mortality, and the composite, as well as the outcomes of 30 day rehospitalization or death, and finally for the days out of hospital and alive adjusted to person-year of time

   1. Days from coronary angiogram performed with IOCM to cardiac surgery (1, 2, 3, etc)
   2. Thakar Acute Renal Failure (ARF) score (1 to 17)
2. To examine the interrelationships between time in days between angiogram and surgery and the ARF Score with the Society of Thoracic Surgery (STS) Risk score for mortality

Methods

Study Design: Retrospective cohort

Subjects: Using the Texas Quality Initiative cardiothoracic surgery database, patients who have recorded one preoperative and at least one postoperative serum creatinine (mg/dl).

Excluded Cases

1. Use of contrast agent other than IOCM with the preoperative angiogram
2. Preoperative use of ventricular assist devices and intraaortic balloon counterpulsation.
3. Operations where there is implantation of mechanical assist devices or cardiac transplant

Measurements:

1. CI-AKI will be assessed by several methods during the period from angiography to cardiac surgery:

   1. Kidney Disease International Global Initiative (KDIGO) as a rise in serum creatinine ≥0.3 mg/dl within 48 hours of surgery or ≥1.5 X baseline serum creatinine within seven days after surgery
   2. Conventional composite CI-AKI definition of ≥25% or ≥0.5 mg/dl rise in serum creatinine from baseline to peak
   3. Conventional singular CI-AKI definition of ≥25% rise in serum creatinine from baseline to peak
   4. Conventional singular CI-AKI definition of ≥0.5 mg/dl rise in serum creatinine from baseline to peak
2. CSA-AKI will be defined by several methods:

   1. Kidney Disease International Global Initiative (KDIGO) as a rise in serum creatinine ≥0.3 mg/dl within 48 hours of surgery or ≥1.5 X baseline serum creatinine within seven days after surgery
   2. Conventional composite derived from CI-AKI definition of ≥25% or ≥0.5 mg/dl rise in serum creatinine from baseline to peak
   3. Conventional singular derived from CI-AKI definition of ≥25% rise in serum creatinine from baseline to peak
   4. Conventional singular derived from CI-AKI definition of ≥0.5 mg/dl rise in serum creatinine from baseline to peak
3. MARCE will be the composite of RRT, myocardial infarction, stroke, heart failure, hospitalizations for cardiac reasons, hospitalization for renal reasons, and death
4. RRT will include at least one session of peritoneal dialysis ultrafiltration, hemodialysis, or other form of extracorporeal blood purification
5. All-cause hospitalization, emergency room, and observation unit visits at 30 days, and one-year will be obtained from the Dallas-Fort Worth Hospital Council Education and Research (DFWHC) connected a regional enterprise master person index (REMPI) database
6. All-cause mortality will be reported as inpatient, 30-day, and one-year
7. Days out of the hospital and alive will be derived as the converse of death and hospitalized days and will be adjusted to 100 PY of time exposure
8. Baseline eGFR will be calculated using the CKD-EPI formula

   GFR = 141 X min(Scr/κ,1)α X max(Scr/κ,1)-1.209 X 0.993Age X 1.018 [if female] X 1.159 [if black]

   Where Scr is serum creatinine (mg/dL), κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1.
9. Clinical factors: age, diabetes, Hb, heart failure, operative variables (bypass time, coronary bypass with valve surgery, on-pump, off-pump) and other predictors of CSA-AKI will be reported in baseline characteristics and considered as candidates for multivariable models

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac surgery with or without cardiac valve surgery
2. At least one baseline and postoperative serum creatinine (mg/dl)

Exclusion Criteria:

1. Use of contrast agent other than IOCM with the preoperative angiogram
2. Preoperative use of ventricular assist devices and intraaortic balloon counterpulsation.
3. Operations where there is implantation of mechanical assist devices or cardiac transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Using the Texas Quality Initiative cardiothoracic surgery database, patients who have recorded one preoperative and at least one baseline and postoperative serum creatinine (mg/dl).
Sampling Method: Non-Probability Sample
Enrollment: 965 (Actual)
Dates: Start 2015-01; Primary Completion 2017-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Contrast-induced acute kidney injury | 7 days
  KDIGO definition
Cardiac surgery associated acute kidney injury | 7 days
  KDIGO definition
Major adverse renal and cardiac events | 30 days
  Composite of need for renal replacement therapy, myocardial infarction, stroke, heart failure, hospitalizations for cardiac reasons, hospitalization for renal reasons, and death

SECONDARY OUTCOMES:
Renal replacement therapy | 30 days
  at least one session of peritoneal dialysis ultrafiltration, hemodialysis, or other form of extracorporeal blood purification
Myocardial Infarction | 30 days
  Myocardial infarction as defined by STS
Stroke | 30 days
  Stroke as defined by STS
Heart failure | 30 days
  Heart failure
Hospitalization for renal reasons | 30 days
  Hospitalization for renal reasons
Hospitalization for cardiac reasons | 30 days
  Hospitalization for cardiac reaons
Death | 30 days
  Death
All-cause hospitalization | 30 days
  All-cause hospitalization, emergency room, and observation unit visits at 30 days, and one-year will be obtained from the Dallas-Fort Worth Hospital Council Education and Research (DFWHC) connected a regional enterprise master person index (REMPI) database
Days out of the hospital and alive | 1 year
  Days out of the hospital and alive will be derived as the converse of death and hospitalized days and will be adjusted to 100 PY of time exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Heart and Vascular Institute, Dallas, Texas, United States

REFERENCES:
- [Background] McCullough PA, Brown JR. Effects of Intra-Arterial and Intravenous Iso-Osmolar Contrast Medium (Iodixanol) on the Risk of Contrast-Induced Acute Kidney Injury: A Meta-Analysis. Cardiorenal Med. 2011;1(4):220-234. doi: 10.1159/000332384. Epub 2011 Oct 4. PMID 22164156
- [Background] Chawla LS, Amdur RL, Shaw AD, Faselis C, Palant CE, Kimmel PL. Association between AKI and long-term renal and cardiovascular outcomes in United States veterans. Clin J Am Soc Nephrol. 2014 Mar;9(3):448-56. doi: 10.2215/CJN.02440213. Epub 2013 Dec 5. PMID 24311708
- [Result] Tecson KM, Brown D, Choi JW, Feghali G, Gonzalez-Stawinski GV, Hamman BL, Hebeler R, Lander SR, Lima B, Potluri S, Schussler JM, Stoler RC, Velasco C, McCullough PA. Major Adverse Renal and Cardiac Events After Coronary Angiography and Cardiac Surgery. Ann Thorac Surg. 2018 Jun;105(6):1724-1730. doi: 10.1016/j.athoracsur.2018.01.010. Epub 2018 Feb 2. PMID 29408241